CLINICAL TRIAL: NCT01717716
Title: Role of Sugars in Solution on Subjective Appetite and Short-term Food Intake in Normal Weight 9-14 Year Old Boys
Brief Title: Sugars-containing Beverage and Food Intake in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Mount Saint Vincent University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Assistant Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: REB 2010-017-001
Record Dates: First submitted 2012-10-23; First posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Childhood Obesity
Keywords: boys; obesity; glucose; sucrose; high-fructose corn syrup-55
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Water; trichlorosucrose; Glucose; Sucrose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Calorie-free control (Experimental): Calorie-free control
  Interventions: Dietary Supplement: water with Sucralose
- HFCS-55 drink (Experimental): HFCS-55 drink
  Interventions: Dietary Supplement: water with HFCS
- Glucose drink (Experimental): Glucose drink
  Interventions: Dietary Supplement: water with glucose
- Sucrose drink (Experimental): Sucrose drink
  Interventions: Dietary Supplement: water with sucrose

INTERVENTIONS:
Dietary Supplement: water with Sucralose
  Arms: Calorie-free control
Dietary Supplement: water with HFCS
  Arms: HFCS-55 drink
Dietary Supplement: water with glucose
  Arms: Glucose drink
Dietary Supplement: water with sucrose
  Arms: Sucrose drink

SUMMARY:
The purpose is to determine the effect of sugars in solution on food intake and subjective appetite in 9- to 14-year-old normal weight boys. The investigators hypothesize that food intake after all sugars-containing solutions will be decreased in comparison to the control solution, with similar reductions in FI between high-fructose corn syrup -55 (HFCS-55) and sucrose. Food intake will be measured 60 minutes after consumption of 50g of HFCS-55, sucrose or glucose, or a control treatment. Subjective appetite will be measured at 15, 30, 45, 60 and 90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, boy, born at full term and normal birth weight

Exclusion Criteria:

* Girl, on restricted diet, taking medication that affect appetite or food intake, have significant learning, behavioral, or emotional difficulties

Ages: 9 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Food intake (kcal) | measured at 60 minutes after the treatment

SECONDARY OUTCOMES:
Subjective appetite (mm) | 0-90 minutes
  Subjective appetite (in mm) by visual analogue scale will be determined at 0, 15, 30, 45, 60 and 90 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Department of Applied Human Nutrition, Bedford, Nova Scotia, Canada